CLINICAL TRIAL: NCT01781897
Title: A Randomized Controlled Trial of Acupuncture to Treat Functional Constipation
Brief Title: Electroacupuncture for the Treatment of Functional Constipation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Guangying Huang, professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011CB505203-1
Record Dates: First submitted 2013-01-23; First posted 2013-02-01 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2014-04

CONDITIONS: Functional Constipation
Keywords: acupuncture; electro-acupuncture
MeSH Terms: interventions — Acupuncture Therapy; mosapride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- mosapride (Active Comparator): mosapride
  Interventions: Drug: mosapride
- Electro-acupuncture (Experimental): Electro-acupuncture
  Interventions: Device: acupuncture
- mosapride + sham acupuncture (Sham Comparator): mosapride + sham acupuncture
  Interventions: Device: acupuncture; Drug: mosapride

INTERVENTIONS:
Device: acupuncture — sterile, disposable needles with a length of 40 mm and a diameter of 0.25 mm (Dongbang® Acupuncture Inc, Korea)
  Other Names: Park true/sham devices
  Arms: Electro-acupuncture; mosapride + sham acupuncture
Drug: mosapride — Mosapride Citrate tablet（5mg），Dainippon Sumitomo pharmaceutical Co.Ltd,Japan
  Other Names: GASMOTIN
  Arms: mosapride; mosapride + sham acupuncture

SUMMARY:
The purpose of this study is to investigate the effect of electroacupuncture on functional constipation.

DETAILED DESCRIPTION:
This study will supply significant evidence for using acupuncture to treat functional constipation(FC), and will help us to identify whether it is a therapeutic effect rather than a placebo effect.

ELIGIBILITY:
Inclusion criteria:

* functional constipation according to the Roman Ⅲ standard;
* aged between 18 and 65 years old

Exclusion criteria:

* unconsciousness, psychosis or can't express subjective symptoms;
* pregnant women or women in lactation period;
* serious diseases of the heart, liver, kidney, and others;
* bleeding disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
number of defecation per week | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohu Xu, Doctor, Principal Investigator — HUST(Huazhong University of Science and Technology) Hospital; Feng Hu, Master, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine
Locations (3):
- China (3):
  - Hospital of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Provincial Hospital of TCM, Wuhan, Hubei
  - Institute of Integrated Traditional Chinese and Western Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei